CLINICAL TRIAL: NCT03435692
Title: Post Operative Analgesia After Pediatric Hip Surgery - PCA, Epidural or Lumbar Plexus Catheter: A Prospective Randomized Control Trial
Brief Title: Post Operative Pain Control After Pediatric Hip Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was exhausted prior to enrolling intended number of patients.
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, David Liston, Assistant Professor, Attending Anesthesiologist, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13144
Record Dates: First submitted 2018-01-30; First posted 2018-02-19 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Hip Surgery; Post Operative Pain Control
MeSH Terms: interventions — Analgesia, Patient-Controlled; Passive Cutaneous Anaphylaxis; Fentanyl; Morphine; Lorazepam; Ondansetron; Diphenhydramine; Acetaminophen; Oxycodone; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lumbar Plexus Catheter (Experimental): Children undergoing pediatric hip surgery will have a lumbar plexus catheter placed (with bolus and continuous infusion of ropivacaine) intraoperatively for perioperative pain control.
  An intraoperative pain protocol will dictate if the patient will receive intravenous fentanyl or morphine. Post operative side effects will be controlled with the administration of ondansetron for nausea and vomiting, diphenhydramine for itching, and lorazepam for muscle spasms. Post operative pain control will be managed with as needed (PRN) morphine and oxycodone as well as scheduled acetaminophen.
  Interventions: Procedure: Lumbar Plexus Catheter; Drug: Fentanyl; Drug: Morphine; Drug: Lorazepam; Drug: Ondansetron; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Oxycodone; Drug: Ropivacaine
- Lumbar Epidural Catheter (Active Comparator): Children undergoing pediatric hip surgery will have an epidural catheter placed (with bolus and continuous infusion of ropivacaine) intraoperatively for perioperative pain control.
  An intraoperative pain protocol will dictate if the patient will receive intravenous fentanyl or morphine. Post operative side effects will be controlled with the administration of ondansetron for nausea and vomiting, diphenhydramine for itching, and lorazepam for muscle spasms. Post operative pain control will be managed with as needed (PRN) morphine and oxycodone as well as scheduled acetaminophen.
  Interventions: Procedure: Lumbar Epidural Catheter; Drug: Fentanyl; Drug: Morphine; Drug: Lorazepam; Drug: Ondansetron; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Oxycodone; Drug: Ropivacaine
- Patient Controlled Analgesia (Active Comparator): Children undergoing pediatric hip surgery will have patient controlled analgesia (with morphine) started in the post anesthesia care unit for post operative pain control.
  An intraoperative pain protocol will dictate if the patient will receive intravenous fentanyl or morphine. Post operative side effects will be controlled with the administration of ondansetron for nausea and vomiting, diphenhydramine for itching, and lorazepam for muscle spasms. Post operative pain control will be managed with as needed (PRN) morphine and oxycodone as well as scheduled acetaminophen.
  Interventions: Procedure: Patient Controlled Analgesia; Drug: Fentanyl; Drug: Morphine; Drug: Lorazepam; Drug: Ondansetron; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: Oxycodone

INTERVENTIONS:
Procedure: Lumbar Plexus Catheter — lumbar plexus catheter placed intraoperatively for perioperative pain control
  Other Names: LPC
  Arms: Lumbar Plexus Catheter
Procedure: Lumbar Epidural Catheter — lumbar epidural catheter placed intraoperatively for perioperative pain control
  Other Names: LEC
  Arms: Lumbar Epidural Catheter
Procedure: Patient Controlled Analgesia — Patient Controlled Analgesia (PCA) was started post operatively for perioperative pain control
  Other Names: PCA
  Arms: Patient Controlled Analgesia
Drug: Fentanyl — Intravenous fentanyl was administered in the operating room for induction of anesthesia. Subsequent doses in the operating room were standardized to be given only for heart rate or blood pressure increases > 20% above baseline and occurring more than 30 minutes after the block if applicable.
Drug: Morphine — In the operating room patients, intravenous morphine was administered if patients had a failed block and standardized to be given only for heart rate or blood pressure increases > 20% above baseline and after fentanyl had been administered. Intravenous Morphine was also administered in the operating room if the patient was randomized to the Patient Controlled Analgesia (PCA) arm of the study. Post operatively intravenous Morphine was administered as needed for severe pain.
Drug: Lorazepam — Intravenous Lorazepam was administered as needed for muscle spasm post operatively.
  Other Names: Ativan
Drug: Ondansetron — Intravenous Ondansetron was administered as needed for nausea and vomiting post operatively.
  Other Names: Zofran
Drug: Diphenhydramine — Intravenous Diphenhydramine was administered as needed for itching postoperatively.
  Other Names: Benadryl
Drug: Acetaminophen — Oral Acetaminophen was administered as needed for pain in the Post-Anesthesia Care Unit (PACU) and then scheduled for 72 hours.
  Other Names: Tylenol
Drug: Oxycodone — Oral Oxycodone was administered as needed for breakthrough pain post operatively.
Drug: Ropivacaine — Intravenous Ropivacaine was administered as part of the initial bolus after placement of the lumbar epidural or lumbar plexus catheter and then as a continuous infusion post operatively.
  Arms: Lumbar Epidural Catheter; Lumbar Plexus Catheter

SUMMARY:
Hip surgery in children is painful and the optimal modality for managing post-operative pain has not been established. This prospective randomized controlled trail compares lumbar plexus catheter (LPC), lumbar epidural catheter (LEC) and continuous patient-controlled analgesia (PCA) with intravenous morphine.

DETAILED DESCRIPTION:
Approximately 1 in 1,000 children born in the US have hip dislocation and 10 in 1,000 have hip subluxation requiring surgical intervention. Pain after major hip surgery in children is severe, yet there is no agreement on the most effective method for pain control. Post-operative pain modalities including lumbar epidural catheters (LEC), lumbar plexus catheters (LPC) and intravenous patient controlled analgesia (IV-PCA) have been described. IV-PCA has historically been the standard of care in spite of its numerous associated side effects. Regional anesthesia modalities have gained popularity because of superior pain control with lower opioid requirements.

In this study, the investigators describe the first prospective randomized controlled trial comparing lumbar plexus catheter to alternatives for post-operative pain management in children after major hip surgery. The investigators hypothesized that LPC would be as safe and efficacious as LEC and IV-PCA with the added advantage of a decreased length of stay. The investigators primary aim was to compare hospital length of stay. Secondary aim was to compare pain scores, opioid consumption and opioid-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing unilateral hip surgery, including pelvic innominate osteotomies, proximal femoral osteotomies, and arthrotomies (for open reduction, loose body removal, labral debridement or labral repair).

Exclusion Criteria:

* History of a previous spine surgery, spina bifida, coagulopathy, skin infection, allergies to study medications (i.e. local anesthetics and opioids), patients taking opioids at the time of enrollment and, those having concurrent procedures distal to the hip.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2011-07-15 (Actual); Primary Completion 2014-07-29 (Actual); Study Completion 2014-07-29 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tredwell SJ. Neonatal screening for hip joint instability. Its clinical and economic relevance. Clin Orthop Relat Res. 1992 Aug;(281):63-8. PMID 1499229
- [Background] Horlocker TT, Kopp SL, Pagnano MW, Hebl JR. Analgesia for total hip and knee arthroplasty: a multimodal pathway featuring peripheral nerve block. J Am Acad Orthop Surg. 2006 Mar;14(3):126-35. doi: 10.5435/00124635-200603000-00003. PMID 16520363
- [Background] Choi PT, Bhandari M, Scott J, Douketis J. Epidural analgesia for pain relief following hip or knee replacement. Cochrane Database Syst Rev. 2003;2003(3):CD003071. doi: 10.1002/14651858.CD003071. PMID 12917945
- [Background] Marino J, Russo J, Kenny M, Herenstein R, Livote E, Chelly JE. Continuous lumbar plexus block for postoperative pain control after total hip arthroplasty. A randomized controlled trial. J Bone Joint Surg Am. 2009 Jan;91(1):29-37. doi: 10.2106/JBJS.H.00079. PMID 19122076
- [Background] Block BM, Liu SS, Rowlingson AJ, Cowan AR, Cowan JA Jr, Wu CL. Efficacy of postoperative epidural analgesia: a meta-analysis. JAMA. 2003 Nov 12;290(18):2455-63. doi: 10.1001/jama.290.18.2455. PMID 14612482

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited at Seattle Children's Hospital main campus location. Recruitment period ran from 7/15/11 to 7/29/14.
Pre-assignment Details: 53 patients were assessed and approached for study eligibility. 10 patients refused to participate and 1 patient did not meet inclusion criteria after initial assessment. 42 patients were enrolled and randomized to study groups.
Groups:
- Lumbar Epidural Catheter: Children undergoing pediatric hip surgery will have an epidural catheter placed (with bolus and continuous infusion of ropivacaine) intraoperatively for perioperative pain control.
  An intraoperative pain protocol will dictate if the patient will receive IV fentanyl or morphine. Post operative side effects will be controlled with the administration of ondansetron for nausea and vomiting, diphenhydramine for itching, and lorazepam for muscle spasms. Post operative pain control will be managed with as needed (PRN) morphine and oxycodone as well as scheduled acetaminophen.
- Lumbar Plexus Catheter: Children undergoing pediatric hip surgery will have a lumbar plexus catheter placed (with bolus and continuous infusion of ropivacaine) intraoperatively for perioperative pain control.
  An intraoperative pain protocol will dictate if the patient will receive IV fentanyl or morphine. Post operative side effects will be controlled with the administration of ondansetron for nausea and vomiting, diphenhydramine for itching, and lorazepam for muscle spasms. Post operative pain control will be managed with PRN morphine and oxycodone as well as scheduled acetaminophen.
- Patient Controlled Analgesia: Children undergoing pediatric hip surgery will have patient controlled analgesia (with morphine) started in the post anesthesia care unit for post operative pain control.
  An intraoperative pain protocol will dictate if the patient will receive IV fentanyl or morphine. Post operative side effects will be controlled with the administration of ondansetron for nausea and vomiting, diphenhydramine for itching, and lorazepam for muscle spasms. Post operative pain control will be managed with PRN morphine and oxycodone as well as scheduled acetaminophen.
Period: Overall Study
Arm/Group | Lumbar Epidural Catheter | Lumbar Plexus Catheter | Patient Controlled Analgesia
Started | 17 | 18 | 7
Completed | 15 (Discontinued intervention (n=2). 1) Lumbar Epidural Catheter (LEC) not working Post-Operative Day (POD) 0, Lumbar Epidural Catheter (LEC) removed and morphine infusion started - patient 1 year old. 2) Lumbar Epidural Catheter (LEC) not working Post-Operative Day (POD) 1, Lumbar Epidural Catheter (LEC) removed and Patient Controlled Analgesia (PCA) started.) | 16 (Discontinued intervention (n=2). 1) Successful lumbar plexus injection, but unable to thread catheter, morphine infusion started (patient 1 year old). 2) Lumbar Plexus Catheter (LPC) catheter (10 cm) not long enough to reach lumbar plexus in patient weighing 136kg, Lumbar Epidural Catheter (LEC) placed instead.) | 7
Not Completed | 2 | 2 | 0
Not completed — Lack of Efficacy | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lumbar Epidural Catheter (< 6 Years Old); Lumbar Epidural Catheter (6 Years and Older): Children undergoing pediatric hip surgery will have an epidural catheter placed (with bolus and continuous infusion of ropivacaine) intraoperatively for perioperative pain control.
- Lumbar Plexus Catheter (< 6 Years Old); Lumbar Plexus Catheter (6 Years and Older): Children undergoing pediatric hip surgery will have a lumbar plexus catheter placed (with bolus and continuous infusion of ropivacaine) intraoperatively for perioperative pain control.
- Patient Controlled Analgesia (6 Years and Older): Children undergoing pediatric hip surgery will have patient controlled analgesia (with morphine) started in the post anesthesia care unit for post operative pain control.
- Total: Total of all reporting groups
Arm/Group | Lumbar Epidural Catheter (< 6 Years Old) | Lumbar Plexus Catheter (< 6 Years Old) | Lumbar Epidural Catheter (6 Years and Older) | Lumbar Plexus Catheter (6 Years and Older) | Patient Controlled Analgesia (6 Years and Older) | Total
Number analyzed (Participants) | 10 | 9 | 7 | 9 | 7 | 42
Age, Customized [Count of Participants; unit: Participants]
  < 6 years old | 10 | 9 | 0 | 0 | 0 | 19
  6 to 18 years old 6 to 18 years old | 0 | 0 | 7 | 9 | 7 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 5 | 3 | 5 | 31
  Male | 0 | 1 | 2 | 6 | 2 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
American Society of Anesthesiologists (ASA) Physical Status Classification System [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) Physical Status Classification System purpose is to assess and communicate a patient's pre-anesthesia medical co-morbidities.
  ASA I is a normal healthy patient. ASA II is a patient with mild systemic disease. ASA III is a patient with severe systemic disease. ASA IV is a patient with severe systemic disease that is a constant threat to life. ASA V is a moribund patient who is not expected to survive without the operation. ASA VI is a declared brain-dead patient whose organs are being removed for donor purposes.
  Participants
    American Society of Anesthesiologists (ASA) Physical Status I | 7 | 6 | 3 | 1 | 4 | 21
    American Society of Anesthesiologists (ASA) Physical Status 2 | 2 | 3 | 3 | 6 | 3 | 17
    American Society of Anesthesiologists (ASA) Physical Status 3 | 1 | 0 | 1 | 2 | 0 | 4
Surgical Approach [Count of Participants; unit: Participants]
  Anterior w/ Osteotomy | 6 | 4 | 2 | 4 | 3 | 19
  Anterior | 2 | 1 | 2 | 4 | 1 | 10
  Lateral w/ Osteotomy | 2 | 4 | 3 | 1 | 3 | 13
Diagnosis [Count of Participants; unit: Participants]
  Femoroacetabular Impingement | 0 | 0 | 4 | 5 | 4 | 13
  Hip Dysplasia | 10 | 9 | 1 | 4 | 1 | 25
  Other | 0 | 0 | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Total hospital length of stay
Time Frame: Through hospital stay, an average of 2-3 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lumbar Epidural Catheter (< 6 Years Old) | Lumbar Plexus Catheter (< 6 Years Old) | Lumbar Epidural Catheter (6 Years and Older) | Lumbar Plexus Catheter (6 Years and Older) | Patient Controlled Analgesia (6 Years and Older)
Number analyzed (Participants) | 10 | 9 | 7 | 9 | 7
days | 1.9 (0.5) | 2 (0.8) | 2.9 (0.8) | 2.5 (1.3) | 3.2 (1.1)

2. Primary Outcome: Maximum Pain Score
Description: Mean of Maximum Pain Score POD 0-2
  Face, Legs, Activity, Cry, Consolability Pain Scale (FLACC) for children 1-3 years of age, Faces Pain Scale - Revised (FPS-R) for children over age 3 and the Numeric scale (0-10) for children over age 7.
  minimum value = 0, maximum value 10 (higher score is worse)
Time Frame: Post-Operative Days 0-2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumbar Epidural Catheter (< 6 Years Old) | Lumbar Plexus Catheter (< 6 Years Old) | Lumbar Epidural Catheter (6 Years and Older) | Lumbar Plexus Catheter (6 Years and Older) | Patient Controlled Analgesia (6 Years and Older)
Number analyzed (Participants) | 10 | 9 | 7 | 9 | 7
score on a scale | 5.5 (0.9) | 4.3 (1.7) | 6.4 (1.7) | 5.5 (1.1) | 6.5 (1.7)

3. Primary Outcome: Total Perioperative Morphine Equivalents
Description: All administered opioids measured as morphine equivalents (mg/kg)
Time Frame: Post-Operative Days 0-2
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Lumbar Epidural Catheter (< 6 Years Old) | Lumbar Plexus Catheter (< 6 Years Old) | Lumbar Epidural Catheter (6 Years and Older) | Lumbar Plexus Catheter (6 Years and Older) | Patient Controlled Analgesia (6 Years and Older)
Number analyzed (Participants) | 10 | 9 | 7 | 9 | 7
mg/kg | 0.54 (0.3) | 0.7 (0.4) | 0.85 (0.4) | 0.83 (0.3) | 2.23 (1.1)

4. Secondary Outcome: Nausea
Description: % of patients with nausea
Time Frame: Post-Operative Days 0-2
Measure: Number; unit: percentage of participants
Arm/Group | Lumbar Epidural Catheter (< 6 Years Old) | Lumbar Plexus Catheter (< 6 Years Old) | Lumbar Epidural Catheter (6 Years and Older) | Lumbar Plexus Catheter (6 Years and Older) | Patient Controlled Analgesia (6 Years and Older)
Number analyzed (Participants) | 10 | 9 | 7 | 9 | 7
percentage of participants | 40 | 33.3 | 71.4 | 55.6 | 71.4

5. Secondary Outcome: Itching
Description: % of patients with itching
Time Frame: Post-Operative Days 0-2
Measure: Number; unit: percentage of participants
Arm/Group | Lumbar Epidural Catheter (< 6 Years Old) | Lumbar Plexus Catheter (< 6 Years Old) | Lumbar Epidural Catheter (6 Years and Older) | Lumbar Plexus Catheter (6 Years and Older) | Patient Controlled Analgesia (6 Years and Older)
Number analyzed (Participants) | 10 | 9 | 7 | 9 | 7
percentage of participants | 40 | 33.3 | 28.6 | 22.2 | 42.9

6. Secondary Outcome: Muscle Spasm
Description: % of patients w/ muscle spasm
Time Frame: Post-Operative days 0-2
Measure: Number; unit: percentage of participants
Arm/Group | Lumbar Epidural Catheter (< 6 Years Old) | Lumbar Plexus Catheter (< 6 Years Old) | Lumbar Epidural Catheter (6 Years and Older) | Lumbar Plexus Catheter (6 Years and Older) | Patient Controlled Analgesia (6 Years and Older)
Number analyzed (Participants) | 10 | 9 | 7 | 9 | 7
percentage of participants | 80 | 55.6 | 100 | 44.4 | 71.4

ADVERSE EVENTS:
Time Frame: Up to 5 days
Description: Adverse event data was collected from the time of enrollment through the participants' study completion. Study completion was defined as when subjects were either discharged from the hospital or removal of the study catheter (lumbar plexus catheter or lumbar epidural catheter) occurred; whichever occurred later. This time period was on average 3 days and no longer than 5 days total.
Arm/Group | Lumbar Epidural Catheter (< 6 Years Old) | Lumbar Plexus Catheter (< 6 Years Old) | Lumbar Epidural Catheter (6 Years and Older) | Lumbar Plexus Catheter (6 Years and Older) | Patient Controlled Analgesia (6 Years and Older)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/7 | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/7 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/7 | 0/9 | 0/7

LIMITATIONS AND CAVEATS:
This study was terminated early because funding was exhausted prior to enrolling intended number of patients. Based on the pre study power analysis we planned to recruit 75 patients; however, we were only able to enroll 42 patients due to limited funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No